CLINICAL TRIAL: NCT06141837
Title: Pseudomonas Aeruginosa Infections Among COVID-19 Patients in Intensive Care Units at Nancy University Hospital During the First Three Epidemic Waves: a Retrospective Study (Pyo-COVID-3)
Brief Title: Pseudomonas Aeruginosa Infections Among COVID-19 Patients in Intensive Care Units at CHRU of Nancy (Pyo-COVID-3)
Acronym: Pyo-COVID-3
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, FLORENTIN Arnaud, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2023PI186
Record Dates: First submitted 2023-11-14; First posted 2023-11-21 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Pseudomonas Aeruginosa; COVID-19
Keywords: ICU infections; antimicrobial resistance
MeSH Terms: conditions — Pseudomonas Infections; COVID-19 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Included: Patient hospitalized between 01/03/20 and 31/05/21 in an intensive care unit of the Nancy University Hospital for at less 48 h for COVID-19 acute respiratory distress syndrome and presenting a positive sample for P. aeruginosa during his stay in the intensive care unit.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No intervention: observational study

SUMMARY:
P. aeruginosa is an opportunistic bacterium known to be responsible for numerous healthcare-associated infections, particularly in intensive care units (ICU). The frequency of these infections seems to have increased during the first waves of the COVID-19 pandemic. Identifying cases of co-infection and secondary infections with P. aeruginosa in patients with COVID-19 would provide a better understanding of the epidemiological evolution and characteristics of infected patients.

Treatment of P. aeruginosa infections requires the use of antibiotics. Antibiotic resistance is a growing problem, with an increase in resistance among P. aeruginosa strains. The misuse of antibiotics to treat patients can accentuate the phenomenon of antibiotic resistance, and failure to take account of resistance revealed by antibiograms can compromise patient recovery. Analysis of bacteriological results and patient medical records would enable a posteriori evaluation of the proper use of antibiotics (choice and adaptation of molecules, doses and duration of prescriptions), and identify any areas for improvement.

The main objective is to describe the evolution of P. aeruginosa infections in ICU patients with COVID-19 during the first 3 waves of COVID-19 (01/03/2020 to 31/05/2021). Secondary objectives are to describe the typology of P. aeruginosa strains identified among included patients (sampling sites and resistance profiles), to assess antibiotic prescriptions for these patients and to describe the relapse rate of included patients with a first P. aeruginosa infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients hospitalized for at least 48 h in an intensive care unit (ICU) at CHRU-Nancy for acute respiratory distress syndrome due to COVID-19.
* Patients hospitalized from 1st March 2020 to 31st May 2021.
* Patient developed an hospital-acquired infection caused by P. aeruginosa during their ICU stay.

Exclusion Criteria:

* Patients <18 years old.
* Patient without COVID-19 at the ICU admission.
* Patients with P. aeruginosa isolated <48 hours following ICU admission.
* Patients who did not want to be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient hospitalized between 01/03/20 and 31/05/21 in an intensive care unit of the Nancy University Hospital for at less 48 h for COVID-19 acute respiratory distress syndrome and developed an hospital-acquired infection caused by P. aeruginosa during their stay in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
P. aeruginosa occurence | From 01 March 2020 to 31 May 2021.
  The occurrence of Pseudomonas aeruginosa infection during the ICU stay of a COVID-19 patient.

SECONDARY OUTCOMES:
P. aeruginosa sample | From 01 March 2020 to 31 May 2021.
  Distribution of different types of samples (respiratory, blood, urine, etc.) positive for P. aeruginosa.
P. aeruginosa resistance | From 01 March 2020 to 31 May 2021.
  The proportion of resistance to the various antibiotics tested on the P. aeruginosa strains identified.
P. aeruginosa antibiotic treatment | From 01 March 2020 to 31 May 2021.
  Compliance of antibiotic prescriptions with reference recommendations is assessed by comparing data from patients' medical records.
P. aeruginosa recurrence | From 01 March 2020 to 31 May 2021.
  Occurrence of a new P. aeruginosa infection.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Florentin, Dr, Principal Investigator — a.florentin@chru-nancy.fr